CLINICAL TRIAL: NCT00169884
Title: The Efficacy of a Cognitive-Behavioural Intervention in Deliberate Self-Harm Patients: A Randomized Controlled Trial Among Adolescents and Young Adults
Brief Title: The Efficacy of a Cognitive-Behavioural Intervention in Deliberate Self-Harm Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2100.0068
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2006-02-01 (Estimated); Status verified 2005-01

CONDITIONS: Self-Injurious Behavior
Keywords: Deliberate Self-Harm,; cognitive-behavioural therapy,; integrative approach
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: cognitive-behavioural therapy

SUMMARY:
The purpose of this study is to evaluate whether the proposed cognitive-behavioural intervention is effective for DSH patients in the age group 15-35 years. In addition, we will examine which elements derived from the theoretical model can explain the efficacy of the intervention.

DETAILED DESCRIPTION:
1. The development of treatment interventions for non-fatal deliberate self-harm (DSH) among young people has received little attention in scientific literature and in mental health care. This is surprising, considering the relatively high rates of hospital-referred DSH among adolescents reported in epidemiological studies (Arensman et al., 1995; Hawton et al., 1997; Hawton et al., 1998; Schmidtke et al., 1996). On the basis of a four-year monitoring study (1989-1992) in the area of Leiden, the average rate of DSH among females aged 15-24 was 179 per 100,000 and for males in this age group the average rate was 91 per 100,000 (Arensman et al., 1995). General population surveys among adolescents show a self-reported life-time prevalence of 2 to 5 percent (Kienhorst et al., 1990; De Wilde et al., 2000). Reports from other European countries indicate an increase of DSH in adolescents and young adults (15-30 years), in particular in young males (Hawton et al., 1997; Schmidtke et al., 1996).

   DSH is operationalized as dysfunctional behaviour associated with a heterogeneity of psychological or psychiatric disorders e.g., affective disorders, anxiety disorders, substance abuse, and eating disorders (Arensman & Kerkhof, 1996; Arensman, 1997; Ellis et al., 1996; Engstroem et al., 1996; Kienhorst et al., 1993). However, a common finding is that depressive symptoms (observer- or self-rated) and major depression appear to be highly prevalent among young DSH patients (Burgess et al., 1998; Goldston et al., 1998; Harrington et al., 1994). In these studies, co-morbidity with other types of psychopathology also appeared to be relatively high.

   The risk of repeated DSH is highest in the first year following an episode of DSH. The repetition rates among young DSH patients vary from 10% (Goldacre & Hawton, 1985) to 27% (Arensman, 1997) in hospital referred DSH patients. Among DSH patients, prevention of the first subsequent repeated episode of DSH is important in order to prevent a pattern of chronic repetition.

   Research findings with regard to risk factors associated with repeated DSH are fairly consistent. Among young DSH patients, those with an increased risk for repeated DSH are characterised by suicidal ideation, depression (Harrington et al., 2000; Hawton et al., 1999), hopelessness (Brent, 1987; Hawton et al., 1999), impulsivity (Kashden et al., 1993), disturbance of autobiographical memory (Evans et al., 1992), problems with peers or other relationships, frequent or chronic stress and problem-solving deficits (De Wilde et al., 2000; Hawton et al., in press; Rudd et al., 1998).

   Despite the fact that many studies report these correlates, the available treatment studies, which merely comprise evaluations of general treatment interventions, often without a randomised controlled design, have not incorporated knowledge about risk factors (Hawton et al., 1998). In addition, existing explanatory and treatment models do not address the heterogeneity of the group of DSH patients. This is surprising, considering the variety of characteristics and problems of DSH patients. So far, most models focus on single psychiatric problems, such as depression or anxiety disorders.

   The aim of this study is to present and test a therapeutic approach for DSH that goes beyond single psychiatric diagnoses and that addresses the heterogeneity of DSH patients. It will combine elements from cognitive-behavioural therapy, problem-solving interventions and Dialectical Behaviour Therapy (DBT), since these approaches fit in with the needs of different DSH patients. Patients in which depressive thoughts and beliefs predominate may especially profit from the elements from cognitive therapy, while patients who primarily experience problems in regulating their emotions may especially profit from the elements from DBT. Patients in whom skills deficits predominate may especially profit from the elements from problem solving interventions. In addition to this combined treatment approach, attention will be given to specific developmental issues that play a role among adolescent DSH patients. Furthermore, knowledge of risk factors for (repetition of) DSH will be incorporated in the treatment.

   The model of the aetiology and maintenance of DSH on which the treatment protocol is based addresses interactions between cognitive, affective, behavioural and interpersonal aspects of DSH. As in other stress-process models, the relationship between vulnerability factors (negative family experiences and biological characteristics), triggering factors, and DSH is mediated by moderating variables (interpersonal problems/lack of social support and individual characteristics: cognitive distortions, affective dysregulation and skills deficits) and mediating variables (negative appraisal, inadequate coping and psychological reactions such as impulsivity). In accordance with Van Praag (1996), we assume that if a person with a marginally functioning serotonergic-system experiences a stressful event he or she is not able to cope with, the production of the stress-hormone cortisol increases, which decreases the level of serotonin. Reduced serotonin activity in the prefrontal cortex as examined by neuroimaging techniques, may be involved in the destabilisation of the regulation of fear, aggression (Van Praag, 1996) and impulsivity (Mann, 1999), since this area of the brain mediates behavioural inhibition. Increased impulsivity may therefore increase the risk of DSH (Van Heeringen, 2001). We assume that in some patients impulsivity and carelessness will be the primary features associated with DSH. In particular, if impulsivity and feelings of hopelessness co-occur, the risk of DSH appears to be high. The recognition of the association between hopelessness and DSH, described here, is in line with the cognitive approach of Williams (2002) stating that over time, among people who perceive they cannot change the stressful situation they are in, despair gradually gains the upper hand and they will show more marked symptoms of depression and hopelessness in particular.The approach as outlined by us, will have advantages compared to approaches based on single psychiatric problems, since it combines the main biological, cognitive, affective, behavioural and interpersonal aspects of DSH.
2. The wide range of problems faced by young people who harm themselves calls for a variety of different treatment strategies, varying from intensive care for those at very high risk of suicide, to brief interventions for the group of patients in whom DSH appears to have been a transient response to temporary difficulties and who have few other problems (Harrington, 2001). One of the most important obstacles to treating DSH patients that may play a role in almost every treatment is compliance (Heard, 2000 in: Hawton and Van Heeringen). Another obstacle in treating DSH patients is the limited availability of research data on effectiveness of therapy for DSH, especially of randomised controlled trials. In the section that follows the most common treatment approaches for DSH will be discussed. Attention will be given to what is known about the effectiveness in terms of reduction of repeated episodes of DSH. Cognitive therapy for DSH patients generally focuses on their tendency to evaluate events and the presence and the future in such a way that this results in the feeling of being entrapped (because of difficulties in coping) and hopelessness (because they have great difficulty in generating positive future events) (Heard, 2000 in: Hawton and van Heeringen). Cognitive and cognitive behavioural therapies directed at cognitive restructuring seem to be promising in successfully treating patients who harm themselves deliberately (Hawton et al., 1998).Given that problem-solving deficits appear to be related to increased risk of self-harm (Orbach et al., 1990), the most commonly used technique for older adolescents is brief problem oriented counselling, which is a form of cognitive therapy. While problem-solving therapy seems to be promising to improve depression, hopelessness and problem-solving skills (Towsend et al., 2001), it is still unclear whether problem-solving therapy can help not only address current problems but also longstanding deficiencies in problem-solving skills. Current research focuses almost exclusively on solving real or hypothetical problems in relationships with other people, yet one of the major issues for suicidal patients is how they can solve the problem of how to gain control over their feelings. Linehan (1993a, 1993b) developed an intensive treatment programme for patients with borderline personality disorder, called Dialectical Behaviour Therapy (DBT). This treatment method focuses on teaching skills that will help people to regulate their emotions and that stress the acceptance of pain and crisis. In a review by Heard (2000 in: Hawton and van Heeringen), in general, a decrease in repeated DSH was found among patients in DBT treatment. Group therapy seems to be promising as a treatment for adolescents who repeatedly harm themselves. However, larger studies are required to assess more accurately the efficacy of this intervention (Wood, Trainor, Rothwell, Moore, Harrington, 2001). No consensus on how to treat DSH medically has been reached yet. As for the psychological treatments, most studies on the efficacy on psychopharmacological treatments are too small to detect significant effects. So far, it appears that the most promising treatments are high doses of Serotonin Specific Reuptake Inhibitors (SSRIs), and, in selected cases atypical neuroleptics. SSRIs are probably the first line medical treatment (Kavoussi et al., 1994). Tricyclics do not seem to be effective for child and adolescent depressions and are toxic in overdose (Harrington, 2001). In conclusion, it can be said that there still remains considerable uncertainty about which type of psychosocial and medical treatments of DSH patients is most effective, inclusion of insufficient numbers of patients in trials being the main limiting factor. However, cognitive-behavioural therapies and problem-solving therapies and DBT seem to be promising. The present study will incorporate elements from cognitive-behavioural therapy, problem-solving interventions and DBT.
3. Study design. The subjects will be randomly allocated to the cognitive-behavioural intervention (experimental group) and routine aftercare (control group), stratified with respect to repetition of DSH and gender.The study subjects are patients aged 15-35 who are referred to the Leiden University Medical Center, to MCH Westeinde (The Hague), or to local centers mental healthcare in Leiden (Rivierduinen)and The Hague (Parnassia PMC), following an act of DSH. DSH patients will be included if they recently have been engaged in an act of DSH including overdoses of medication, ingestion of chemical substances and self-inflicted injuries according to the definition which is used in the WHO/Euro Multicentre Study on parasuicide: "An act with non-fatal outcome in which an individual deliberately initiates a non-habitual behaviour, that without intervention from others will cause self-harm, or deliberately ingests a substance in excess of the prescribed or generally recognised dosage, and which is aimed at realising changes that the person desires via the actual or expected physical consequences" (Platt et al., 1992). DSH patients with severe psychiatric disorders requiring intensive long-term psychiatric treatment will be excluded.

ELIGIBILITY:
Inclusion Criteria:

DSH patients will be included if they recently have been engaged in an act of DSH including overdoses of medication, ingestion of chemical substances and self-inflicted injuries according to the definition which is used in the WHO/Euro Multicentre Study on parasuicide: "An act with non-fatal outcome in which an individual deliberately initiates a non-habitual behaviour, that without intervention from others will cause self-harm, or deliberately ingests a substance in excess of the prescribed or generally recognised dosage, and which is aimed at realising changes that the person desires via the actual or expected physical consequences" (Platt et al., 1992). In addition, only DSH patients aged 15-35 will be included.

Exclusion Criteria:

DSH patients with severe psychiatric disorders requiring intensive long-term psychiatric treatment, such as schizophrenia, will be excluded.

Ages: 15 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120
Dates: Start 2002-03; Study Completion 2007-03

PRIMARY OUTCOMES:
repetition of DSH

SECONDARY OUTCOMES:
psychiatric diagnosis, depression, hopelessness, suicidal intent, suicidal cognitions, self-concept, (cognitive) coping, emotion regulation difficulties, impulsivity, social support, hostility, personality disorder related beliefs and attachment style.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Spinhoven, prof. dr., Study Chair — Leiden University, department of clinical psychology; Nadia Garnefski, dr., Study Director — Leiden University department of clinical psychology; Nadja Slee, MSc, Principal Investigator — Leiden University department of clinical psychology; Ella Arensman, dr., Study Director — National Suicide Research Foundation, Cork
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - MCH Westeinde, The Hague

REFERENCES:
- See also: Related Info — http://www.fsw.leidenuniv.nl